CLINICAL TRIAL: NCT04637373
Title: Hysteroscopy Assisted Suction Curettage for Early Pregnancy Loss: Does it Reduce Retained Products of Conception and Postoperative Intrauterine Adhesions?
Brief Title: Hysteroscopy Assisted Suction Curettage for Early Pregnancy Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Omer Moore, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0178-19-ASF
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Retained Products of Conception; Intrauterine Adhesion
Keywords: intrauterine adhesions; Hysteroscopy; Retained Products of Conception
MeSH Terms: conditions — Gynatresia | interventions — Hysteroscopy

STUDY DESIGN:
Intervention Model Description: This prospective descriptive study is taking place in a single university affiliated medical center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the group (Experimental): Women aged 18-40 years who admit to the gynecology emergency department at our institution with early miscarriage up to 12 weeks and 6 days of gestation, and choose surgical evacuation over medical treatment, are having Hysteroscopy assisted suction curettage as detailed previously. retained products of conception found at the end of the procedure, and intrauterine adhesions found on follow up are compared to the data in the literature.
  Interventions: Diagnostic Test: Hysteroscopy

INTERVENTIONS:
Diagnostic Test: Hysteroscopy — adding Hysteroscopy before and after suction curettage for early missed abortion to define the wall of implantation and look for retained products of conception

SUMMARY:
Retained products of conception (RPOC) and intrauterine adhesions (IUA) may occur following suction curettage for early miscarriage and cause secondary infertility, recurrent pregnancy loss and pregnancy complications. The aim of this study is to investigate whether adding hysteroscopy to suction curettage reduces the rates of RPOC and IUA.

DETAILED DESCRIPTION:
This is a descriptive, prospective study. Women aged 18-40 years admitted for surgical evacuation in cases of early missed abortion in a single university affiliated medical center are being recruited. All procedures performed under general anesthesia following cervical ripening with vaginal Misoprostol.

Before the evacuation, a diagnostic hysteroscopy was performed to identify the pregnancy's implantation wall. Subsequently, ultrasound guided suction and curettage directed to the implantation wall is done. Finally, the uterine cavity is evaluated by hysteroscopy for RPOC. Participants are scheduled for follow-up diagnostic office hysteroscopy 2 months after termination of pregnancy for assessment of IUA and RPOC. However, due to restrictions on elective surgical procedures brought on by the Covid-19 pandemic, the follow-up hysteroscopy examination was postponed until 5 to 6 months after termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years who were admitted to the gynecology emergency department at our institution with early miscarriage up to 12 weeks and 6 days of gestation, and choose surgical evacuation over medical treatment

Exclusion Criteria:

* incomplete and complete abortions, gestational age>13 weeks of gestation, suspected molar pregnancy and patients' contraindications for general anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the occurrence of Retained products of conception following suction curettage. | at the end of suction curettage procedure

SECONDARY OUTCOMES:
the occurrence of intra uterine adhesions following targeted suction curettage | on follow-up office hysteroscopy, 5-6 months after the primary procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Yes, going to publish, not deciced on which paper yet